CLINICAL TRIAL: NCT00307866
Title: A Prospective, Multicenter, Phase III b Clinical Study to Evaluate the Effectiveness of Unenhanced and SH U 555A (Resovist) Enhanced MRI, Compared to Contrast-Enhanced Dual-Phase Spiral CT in Assessing the Correct Final Therapy-Deciding Diagnosis, in Patients With Primary or Secondary Hepatic Malignancies.
Brief Title: Identification of Hepatic Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 90956; 304668
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Hepatic Neoplasms
Keywords: Known or suspected focal liver lesions detected by spiral CT
MeSH Terms: conditions — Liver Neoplasms | interventions — ferumoxides

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Procedure: Resovist (BAY86-4884, SH U 555 A)

INTERVENTIONS:
Procedure: Resovist (BAY86-4884, SH U 555 A) — Single bolus injection, followed by MRI

SUMMARY:
Patients with suspicion of primary or secondary hepatic malignancy in whom a radiological examination is needed in order to decide on the most appropriate treatment.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Present with suspicion of primary or secondary hepatic malignancy in whom a radiological examination is needed in order to decide on the most appropriate treatment. There should not be more than five liver lesions on type visualized on CT.

   The patient should be in a condition that allows subsequent treatment.
2. Be willing and able to continue study participation following administration of SH U 555 A to ensure completion of all procedures and observations required by the trial protocol.
3. Sign and date fully informed consent prior to entry into the study.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients weighing less than 35 kg.
* Patients who have received any investigational drug within the 30 days prior to entering this study.
* Patients who have previously entered this study or any other study performed with SH U 555 A.
* Women who are pregnant or who are of childbearing potential and have not had a negative urine pregnancy test immediately prior to the administration of SH U 555 A. The urine pregnancy test should be performed in accordance with the manufacturer's recommendations.
* Lactating women.
* Patients who have any contraindication to MRI examination.
* Patients who have received any contrast material in the 24 hours prior to SH U 555 A injection, or who are scheduled to receive any contrast material within 24 hours afterwards. (In the case of any liver specific agent (e.g. MnDPDP, SPIOs, Gd-BOPTA) this will be extended to 14 days prior to the study).
* Patients who have received Lipiodol contrast material at any time in the past or are scheduled to receive this during the study period.
* Patients who are clinically unstable and whose clinical course during the observation period is unpredictable (e.g. due to previous surgery).
* Patients scheduled for liver biopsy within 24 hours, or who had a biopsy within the 24 hours prior to planned SH U 555 A injection.
* Patients who are scheduled for, or are likely to require, surgery within 24 hours after SH U 555 A injection.
* Patients with a history of anaphylactoid or anaphylactic reaction to any allergen including drugs and contrast agents.
* Patients with known hypersensitivity to any of the ingredients of SH U 555 A.
* Patients with already clear op-indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2001-04; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
To assess the proportion of correct final, therapy deciding diagnosis based on unenhanced plus SH U 555 A enhanced MR imaging compared to contrast-enhanced dual-phase spiral CT.

SECONDARY OUTCOMES:
To assess the number, size , location and character of liver lesions.
To assess the diagnostic confidence of MRI and CT.
To assess the proportion of changed therapeutical decisions.
To assess sensitivity and specificity of MRI and CT.
To assess safety and tolerability of SH U 555 A administration.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- Italy (17):
  - Bari, BA
  - Bologna, BO
  - Brescia, BS
  - Florence, FI
  - Genova, GE
  - Milan, MI
  - Palermo, PA
  - Pisa, PI
  - Roma, Roma
  - Sassari, SS
  - Torino, TO
  - Trieste, TS
  - Verona, VE
  - Chieti
  - L’Aquila
  - Roma
  - Udine